CLINICAL TRIAL: NCT04512560
Title: Structured Remote Surgical Coaching to Improve Operative Performance in Laparoscopic Cholecystectomy: a Multicenter Randomized Control Trial
Brief Title: Structured Remote Surgical Coaching to Improve Operative Performance in Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Boris Zevin (Other)
Responsible Party: Sponsor-Investigator, Dr. Boris Zevin, Assistant Professor & Medical Education Scholar, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SURG-497-20
Record Dates: First submitted 2020-03-31; First posted 2020-08-13 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-07

CONDITIONS: Education; Coaching; Surgical; Laparoscopic; Cholecystectomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Technical skills and technical errors will be assessed by a trainer rater blinded to the participant's group allocation and level of training.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Structured Remote Surgical Coaching (Experimental): Participants randomized to the intervention group will participate in a 3-month SRSC program in addition to CST. Participants will be asked to provide a video recording of a laparoscopic cholecystectomy that they performed as a primary surgeon prior to the coaching session. Each coach will review the video recording and will identify key themes for discussion. Coaching sessions will be structured using the modified PRACTICE model, will be conducted outside of the clinical environment, and will employ facilitative coaching methods to encourage participants to define specific intra-operative problems and conceptually troubleshoot various solutions.
  Interventions: Behavioral: Surgical Training using Structured Remote Surgical Coaching in addition to Conventional Surgical Training
- Conventional Surgical Training (Active Comparator): Participants randomized to the control group will continue of their usual general surgery residency training including attending scheduled teaching sessions, and continuing with assigned responsibilities on the ward and in the OR.
  Interventions: Behavioral: Surgical Training using Conventional Training Program

INTERVENTIONS:
Behavioral: Surgical Training using Structured Remote Surgical Coaching in addition to Conventional Surgical Training — General surgery residents (PGY 1-5) will provide a video recording of a laparoscopic cholecystectomy that they performed as a primary surgeon. The coach will identify key moments or themes for discussion on how to improve technical skills and reduce intra-operative errors during five, 30-45 minute remote coaching sessions .
  Arms: Structured Remote Surgical Coaching
Behavioral: Surgical Training using Conventional Training Program — General surgery residents (PGY 1-5) will continue their usual residency training.
  Arms: Conventional Surgical Training

SUMMARY:
Surgical coaching, defined as a constructive relationship that provides objective feedback to individuals about a broad range of factors influencing operative performance, is a key strategy for integrating adult learning theory into the traditionally didactic arena of surgical education. It is gaining momentum as an area of potential growth and innovation, and may become a more meaningful method of ongoing professional development for practicing surgeons. Effective coaching interactions encourage discussion, provide feedback, affirm positive beliefs and challenge pre-existing assumptions. The effectiveness and uptake of coaching interventions in surgery can be influenced by the identity of the coach, and cultural or individual surgeon attitudes.

Surgical coaching has been linked to improvements in technical and procedural skills in both simulated and clinical environments. In 2015, a systematic review of surgical coaching showed a positive impact of surgical coaching interventions on learners' perceptions and attitudes, their technical and nontechnical skills, and their performance measures.

The investigators propose to conduct a multicenter randomized controlled trial of structured remote surgical coaching (SRSC) versus conventional surgical training for laparoscopic cholecystectomy performed by surgery residents at three institutions, in Canada and Australia, to not only provide additional evidence in support of validity and generalizability of a structured surgical coaching intervention for surgery trainees, but also to demonstrate improvement in accuracy of self-assessment of operative performance and the feasibility of remote coaching.

DETAILED DESCRIPTION:
OBJECTIVES: To compare the effects of adding a structured remote surgical coaching (SRSC) program to conventional surgery training (CST) versus conventional surgery training (CST) alone on general surgery residents' (1) technical performance, (2) technical errors, and (3) accuracy of self-assessment for a laparoscopic cholecystectomy procedure. Feasibility of conducting remote coaching across different times zones and continents will also be explored.

Hypothesis 1: Participation in a SRSC program will result in superior technical skills and fewer technical errors committed during a laparoscopic cholecystectomy as compared to CST.

Hypothesis 2: Participation in a SRSC program will result in a more accurate self-assessment of participants' technical skills as compared to CST.

Hypothesis 3: It will be feasible to coach surgery residents remotely across different time zones and continents.

STUDY DESIGN AND SETTING:

The investigators will conduct a multicenter randomized controlled trial with study participants randomized 1:1 into intervention (SRSC+CST) and control groups (CST). The investigators will use blocked randomization with a block size of 4 and allocation ratio of 1:1 to ensure equal participant distribution over the 24 month continuous recruitment period.

STUDY PARTICIPANTS AND RECRUITMENT:

The investigators will recruit general surgery residents (PGY 1-5) as study participants. Any resident who routinely performs components of a laparoscopic cholecystectomy as a primary surgeon (under supervision) and is rotating on a general surgery service will be invited to participate.

STRUCTURED REMOTE SURGICAL COACHING (SRSC) PROGRAM (INTERVENTION):

Participants randomized to the intervention group will participate in a 3-month SRSC program in addition to CST. They will view a standardized 10-minute video presentation, which will explain the concept of surgical coaching and the purpose of the SRSC program. Surgical coaches will provide structured remote surgical coaching. Credentials and qualifications of each of the coaches are described below (Research Team). Zoom web-conferencing platform (https://zoom.us) will be used for remote coaching. Participants will be asked to provide a video recording of a laparoscopic cholecystectomy that they performed as a primary surgeon prior to the coaching session. Each coach will review the video recording and will identify key themes for discussion. Coaching sessions will be structured using the modified PRACTICE model, will be conducted outside of the clinical environment, and will employ facilitative coaching methods to encourage participants to define specific intra-operative problems and conceptually troubleshoot various solutions. Key observations and discussion points for each session will be recorded in a coaching template. Coaching sessions will be planned to be administered on a bi-weekly basis; however, variability may occur to accommodate residents operating schedule and exposure. The expectation is for each participant to complete three to four coaching sessions each lasting 30-45 minutes.

CONVENTIONAL SURGICAL TRAINING (CONTROL):

Participants randomized to the control group will continue of their usual general surgery residency training including attending scheduled teaching sessions, and continuing with assigned responsibilities on the ward and in the OR. Participants will be asked to record videos of 5 consecutive laparoscopic cholecystectomy procedures that they performed as a primary surgeon during a 3-month period to mimic the duration of exposure in the intervention group.

DEMOGRAPHIC DATA:

The investigators will collect age, sex, post-graduate year of training, handedness, number of basic, intermediate and advanced laparoscopic cases performed as a primary surgeon or assisted before and during the study.

PRIMARY OUTCOME MEASURES:

The investigators will measure technical performance during a laparoscopic cholecystectomy as the primary outcome. Two assessment scales will be used: the Global Operative Assessment of Laparoscopic Skills (GOALS) scale and the Generic Error Rating Tool (GERT) for errors in laparoscopic surgery.

SECONDARY OUTCOME MEASURES:

The investigators will explore, using a post-study questionnaire, the subjective perception of the usefulness of the SRSC program and challenges with remote coaching as the secondary outcome. The investigators will also collect feasibility data including duration of time spent on video review, preparation for the coaching session, and conduct of the session by the coach. Participant self-assessment data for their technical performance at baseline and upon the completion of the study will also be collected.

BASELINE AND POST-INTERVENTION ASSESSMENT:

The 1st and 5th submitted video recording for each study participant will be assessed by a trained rater, blinded to the group allocation and training level of participant, for technical skill and errors using GOALS and GERT scales, respectively. Participants will self-assess their technical performance with the GOALS scale.

SAMPLE SIZE:

Using clinically relevant effect size of 1.25 and 1:1 allocation ratio for groups, a minimum of 9 participants will be required per group to achieve a power of 0.8 and alpha of 0.05. The investigators will aim to recruit a total of 24 participants (12 per group) to account for possible participant dropout. An interim analysis will be performed once 9 participants have been recruited per group. Recruitment will continue until completion of the interim analysis.

DATA ANALYSIS:

The investigators will perform descriptive statistical analysis and will assess the normality of data distribution using the Shapiro-Wilk test. For continuous variables with normal distribution, the investigators will use a t-test for independent samples for between group comparisons, and a paired t-test for within group comparisons. For continuous variables with skewed distribution, the investigators will use the Mann-Whitney U test for between group comparisons, and the Wilcoxon rank sign tests for within group comparisons. The investigators will compare categorical data using the Fisher exact test. The investigators will use Spearman correlations to examine the correlation between self-assessment scores and blinded rater scores.

ELIGIBILITY:
Inclusion Criteria:

* General surgery residents (PGY 1-5) who routinely perform components of laparoscopic cholecystectomy as a primary surgeon (under supervision).

Exclusion Criteria:

* Individuals with injuries that preclude performance in the operating room will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Skill set during performance of a laparoscopic cholecystectomy in the operating room | 90 days
  Technical skills during a laparoscopic cholecystectomy in the operating room will be one of the primary outcomes for this study. The Global Operative Assessment of Laparoscopic Skills (GOALS) scale will be used to measure this outcome.
Technical errors made during a laparoscopic cholecystectomy in the operating room | 90 days
  Technical errors during a laparoscopic cholecystectomy in the operating room will be one of the primary outcomes for this study. The Generic Error Rating Tool (GERT) will be used to measure this outcome.

SECONDARY OUTCOMES:
Subjective assessment of the usefulness of SRSC program | 90 days
  A post-study questionnaire will be administered to participants in the intervention group to assess their subjective perception of the usefulness of the SRSC program and challenges that they encountered with remote coaching.
  A scale for Perception of Usefulness will be used in this post-study questionnaire with a minimum value of 1 indicating not useful at all and a maximum value of 10 indicating very useful.
Accuracy of self-assessment | 90 days
  Participants' self-assessment scores for technical skill will be compared to the scores assigned by a trained, blinded rater to determine if SRSC improves accuracy of self-assessment

CONTACTS AND LOCATIONS:
Overall Officials: Boris Zevin, MD, Principal Investigator — Queen's University
Locations (1):
- Queen's University, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No